CLINICAL TRIAL: NCT02537626
Title: An Evaluation of the Effect of the Erchonia ALS on Alzheimer's Disease
Brief Title: An Evaluation of Low Level Laser Light Therapy on Improving the Symptoms of Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC_AD_001
Record Dates: First submitted 2015-08-27; First posted 2015-09-01 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erchonia ALS Laser (Active Comparator): The Erchonia ALS Laser is a mains powered variable hertz laser device made up of five independent red laser diodes mounted in scanner devices and positioned equidistant from each other. Each scanner emits 7.5 milliwatts (mW) ± 1.0 mW 640 nanometers (nm) with a tolerance of ±10 nm of red laser light.
  Interventions: Device: Erchonia ALS Laser
- Placebo Laser (Placebo Comparator): The Placebo Laser is identical in appearance and operation to the Erchonia ALS Laser but does not emit any therapeutic light.
  Interventions: Device: Placebo Laser

INTERVENTIONS:
Device: Erchonia ALS Laser — The Erchonia ALS Laser is administered to the subject's frontal cortex, temporal regions and base of the skull 8 times across 4 consecutive weeks, 2 times each week, for 10 minutes of treatment time per administration. The total energy delivered to the subject per procedure administration is 22.5 joules.
  Arms: Erchonia ALS Laser
Device: Placebo Laser — The Placebo Laser is administered to the subject's frontal cortex, temporal regions and base of the skull 8 times across 4 consecutive weeks, 2 times each week, for 10 minutes of treatment time per administration. There is no energy delivered to the subject.
  Arms: Placebo Laser

SUMMARY:
This study evaluates the effect of applying low level laser light therapy to individuals with mild to moderate Alzheimer's disease to see if it may improve their memory, thinking and behaviors. Half of the participants will receive the real treatment with the laser device and the other half of the participants will receive a placebo treatment (not active laser).

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a progressive type of dementia that causes problems with memory, thinking and behavior that gradually worsen over time. With an aging population, AD is an escalating problem, currently affecting an estimated 35 million people worldwide, with this number expected to grow to 65 million by 2030 and over 115 million by 2050. It is the sixth leading cause of death in the United States.

AD is a fatal degenerative disease of the brain that causes brain cells to die which as a result causes the memory failure, personality changes, problems carrying out daily activities and other symptoms associated with AD. AD is thought to be caused by an excess of beta amyloid (β-amyloid), a sticky protein in the brain that forms amyloid plaques and tangles that accumulate over time, and are associated with significant loss of neurons and synaptic activity in the brain.

Patients with AD typically first present with impaired memory and language dysfunction, with visuospatial dysfunction, impaired ability with calculations and complex tasks, behavioral and/or psychiatric symptoms developing as the disease progresses. The most common signs and symptoms of AD as the disease progresses are: memory loss that disrupts daily life, challenges in planning or solving problems, difficulty completing familiar home, work or leisure tasks, confusion with time or place, difficulty understanding visual images and spatial relationships, new problems with words in speaking or writing, misplacing things and losing the ability to retrace steps, decreased or poor judgment, withdrawal from work or social activities, changes in mood, personality and behavior.

There is presently no cure for Alzheimer's disease or its progression. Current available treatments can help to lessen or stabilize symptoms for a limited period of time. The FDA has approved two types of medications to treat the cognitive symptoms (memory loss, confusion, and problems with thinking and reasoning) of AD: cholinesterase inhibitors such as Aricept, Exelon, Razadyne, Cognex and memantine (Namenda). Side effects include nausea, dizziness, confusion, vomiting, headache, loss of appetite, constipation, increased frequency of bowel movements, and possible liver damage. Current alternative treatments include Vitamin E.

There are no medications approved specifically to treat behavioral and psychiatric AD symptoms. However, antidepressants; anxiolytics and antipsychotics are sometimes prescribed.

As currently available treatments for AD are minimal and of limited short-term effectiveness in mild symptom management at best, and have potentially serious associated side-effects, low level laser therapy is being evaluated in this study as a simple, non-invasive side-effect free alternate means of improving cognition and behavior symptoms in patients with mild to moderate AD.

The underlying condition of AD is the degeneration and death of nerve cells responsible for memory and cognition with identified genetic contributions. Application of low level laser therapy (LLLT), with its coherent emission of photons, has been shown to modulate cellular metabolism and alter the transcription factors responsible for gene expression to produce cell regeneration translating to a beneficial clinical effect. It is therefore hypothesized that through this mechanism, application of LLLT to individuals with AD will effect improvement in the expression of symptoms of AD. Prior Erchonia Corporation LLLT trials have shown beneficial clinical effects for other neurodegenerative and neurodevelopment disorders such as Parkinson's Disease and Autism Spectrum Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient AD individual with consistent, reliable caregiver willing and able to participate as needed for the duration of the study
* Subject satisfies the Diagnostic and Statistical Manual Of Mental Disorders. 5th Edition (DSM-V) Criteria For Major Neurocognitive Disorder (NCD) Due To Alzheimer's Disease
* Mini-Mental Status Examination (MMSE) score of > 11 to < 26
* Hachinski ischemic score of ≤ 4
* The subject/study partner agrees to report any changes in medication use to the investigator throughout study duration
* 50 to 85 years of age, inclusive
* Subject is ambulatory with or without aid
* Vision and hearing sufficient to comply with testing
* Normal cognitive and social functioning prior to onset of dementia
* Female subjects of child-bearing potential are willing and able to use acceptable means of contraception throughout study participation.
* English speaking subject and study partner

Exclusion Criteria:

* AD individual residing in an inpatient care facility, such as a nursing home
* Likelihood, according to clinical judgment, of being transferred to an inpatient care facility within 6 months
* Life expectancy is less than 6 months
* Non-Alzheimer primary dementia or neurodegenerative disease other than AD, including: vascular dementia; Lewy body dementia; fronto-temporal dementia; multi-infarct dementia; vitamin B-12 deficiency; hypothyroidism; Huntington's Disease; Parkinson's Disease; normal pressure hydrocephalus; cognitive dysfunction due to cerebral damage resulting from a lack of oxygen, a brain injury; cerebral tumor
* Autoimmune disorder, such as HIV, Chronic Fatigue Syndrome and fibromyalgia that in the opinion of the investigator is significant enough to affect the subject's ability to take part in all of the requirements of study participation
* Active cancer or treatment for cancer within the last 6 months
* Unstable cardiac disease, such as a recent cardiac arrhythmias (including atrial fibrillation, ventricular fibrillation and irregular atrial-ventricular conduction time), or recent congestive heart failure, or recent myocardial infarction
* Uncontrolled diabetes
* Known or diagnosed major depressive disorder, schizophrenia, or other significant psychotic disorders, bipolar disorder, or substance (including alcohol and/or drug) related disorders that in the opinion of the investigator may interfere with or affect study outcome evaluation; including hospitalization for psychiatric disturbances within the past 2 years
* Total score of 20 or greater on the Geriatric Depression Scale
* Any other advanced, severe, progressive, unstable and/or uncontrolled systemic disease or illness of any type that in the opinion of the investigator may interfere with study procedure administration and efficacy assessment
* Active infection, wound or other external trauma to the areas to be treated with the laser
* Medical, physical, or other contraindications for, or sensitivity to, light therapy
* Subject is presently pregnant, breast feeding or attempting or planning to attempt to become pregnant during the course of the study participation time frame
* Participation in a research study within the past 30 days
* Subject is not ambulatory

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) Score | 4 months
  The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog) is a validated psychometric instrument to evaluate the following aspects of cognitive function: memory, attention, reasoning, language, orientation, ideational praxis and constructional praxis. Scores on the ADAS-cog range from 0-70 with higher scores indicating greater impairment. Therefore, a decrease in the ADAS-cog score from baseline to study endpoint indicates improved cognitive functioning and is positive for study success; whereas an increase in the ADAS-cog score from baseline to study endpoint reflects potential cognitive deterioration and is negative for study success. The minimal clinical important difference (MCID) on the ADAS-cog has been established as a 4 point change (decrease).
Alzheimer's Disease Co-Operative Study-Activities of Daily Living Inventory (ADCS-ADL) | 4 months
  The Alzheimer's Disease Co-Operative Study-Activities of Daily Living Inventory (ADCS-ADL) is a validated tool to assess instrumental and basic activities of daily living (i.e. functional performance) of AD based on a structured interview of the study partner. Scores on the ADCS-ADL range from 0-78 with lower scores indicating greater impairment; Therefore, an increase in the ADCS-ADL score from baseline to study endpoint indicates improved functioning and is positive for study success; whereas a decrease in the ADCS-ADL score from baseline to study endpoint reflects potential functional deterioration and is negative for study success. The minimal clinical important difference (MCID) on the ADAS-ADL has been established as a 2 point change (increase - improvement).

SECONDARY OUTCOMES:
Mini Mental State Examination (MMSE) | 4 months
  The Mini Mental State Examination (MMSE) tool evaluates five areas of cognitive function: orientation, registration, attention and calculation, recall and language. It is an 11-item tool with a maximum attainable score of 30. A total score of 23 or lower indicates cognitive impairment.
  Lower scores indicate progressively greater impairment. Therefore, an increase in the MMSE score from baseline to study endpoint indicates improved cognition and is positive for study success; whereas a decrease in the MMSE score from baseline to study endpoint reflects potential cognitive deterioration and is negative for study success.
Study Partner Satisfaction With Overall Outcome Rating | 4 months
  The subject's study partner is asked to indicate how satisfied he or she is with any change observed in the subject's day-to-day functioning following the study procedure administration phase. Responses are recorded on a 5-point scale from 'Very Satisfied' to 'Not at All Satisfied'. Higher ratings indicate greater satisfaction with the study outcome and are positive for study success. Lower ratings indicate lesser satisfaction with the study outcome and are negative for study success

CONTACTS AND LOCATIONS:
Overall Officials: Leon Morales-Quezada, MD, Principal Investigator — Neocemod; Andrew Campbell, MD, Principal Investigator — Pruebas Clinicas
Locations (2):
- Mexico (2):
  - Pruebas Clinicas, Zapopan, Jalisco
  - Neocemod, La Plazuela, Pocitos AGS

IPD SHARING:
Plan to Share IPD: No